CLINICAL TRIAL: NCT04023149
Title: Short-term Efficacy of Interleukin-2 Gargle Combined With Systemic Use of Glucocorticoids in the Treatment of Oral Mucosal Lesion in Pemphigus Vulgaris: a Randomized, Controlled, Double-blind, Multicenter Clinical Study
Brief Title: Efficacy of Interleukin-2 Gargle in the Treatment of Oral Mucosa Lesion in Pemphigus Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Qianjin Lu, MD, PhD, Professor and Director, Dept. of Dermatology, The Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPOEMS201903
Record Dates: First submitted 2019-07-03; First posted 2019-07-17 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Pemphigus Vulgaris
Keywords: pemphigus vulgaris; oral mucosal lesion; interleukin-2
MeSH Terms: conditions — Pemphigus | interventions — aldesleukin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients will receive rhIL-2 solution oral gargle twice per day (2 million units of rhIL-2 dissolved in 5ml normal saline for each dose, garble for 3 minutes) and continue for 3 weeks. A standard dose of glucocorticoids (mucosal-dominant PV: prednisone 0.5 mg/kg/d, moderate mucocutaneous PV: prednisone 0.75 mg/kg/d) will be applied at the same time.
  Interventions: Drug: recombinant human interleukin-2 (rhIL-2)
- control group (Placebo Comparator): Patients will receive placebo solution oral gargle twice per day (5ml for each dose, garble for 3 minutes) and continue for 3 weeks. A standard dose of glucocorticoids (mucosal-dominant PV: prednisone 0.5 mg/kg/d, moderate mucocutaneous PV: prednisone 0.75 mg/kg/d) will be applied at the same time.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: recombinant human interleukin-2 (rhIL-2) — Drug: rhIL-2; Pharmaceutical form: solution; Route of administration: oral gargle.
  Arms: experimental group
Drug: placebo — Drug: placebo; Pharmaceutical form: solution; Route of administration: oral gargle.
  Arms: control group

SUMMARY:
This clinical study will test the short-term efficacy of interleukin-2 gargle combined with systemic use of glucocorticoids in the treatment of oral mucosal lesions in mucosal-dominant pemphigus vulgaris and moderate mucocutaneous pemphigus vulgaris.

DETAILED DESCRIPTION:
Backgrounds: Pemphigus vulgaris (PV) is a life-threatening autoimmune bullous skin disease characterized by blisters or bullae on the skin and mucosal membranes. The formation of painful erosion surface after rupture of blisters may result in infection, haemorrhage and even electrolyte imbalance due to excessive water loss. PV can be divided into two types: mucocutaneous PV and mucosal-dominant PV. Patients with mucocutaneous PV not only suffer from severe mucosal damage but also general skin lesions, while slight or no skin lesions involved in patients with mucosal-dominant PV. Oral mucosal damage occurred 3 months to 1 year before skin lesions in about 60% of PV patients. The most common involving parts of the oral mucosa are pars buccalis and oropharynx, presenting with persistent and painful erosion or ulceration, which leads to difficulty in feeding and aggravates the electrolyte imbalance.

Glucocorticoid is the main treatment strategy of PV. Besides the blisters and erosion, complications of long-term use of glucocorticoid are also the death causes of PV patients, such as osteoporosis, hyperglycemia, hypertension, hypokalemia, femoral head necrosis, peptic ulcer, and infection. Many patients have gotten remission from the standard application of glucocorticoids, Immunosuppressants and biological agent. However, there is still a part of patients that are insensitive to these drugs or intolerant the side effects of corticosteroids. Even for those steroid-sensitive patients, the healing of oral mucosa often takes a long course, lasting from weeks to months, which has a serious impact on the quality of life. It is a critical problem to develop novel therapeutics to accelerate the healing of oral mucosa.

Recombinant human interleukin-2 (rhIL-2) is an immunomodulator agent commonly used in the treatment of patients with tumours. The safety and efficacy of low dose rhIL-2 have been demonstrated in the treatment of type I diabetes, systemic lupus erythematosus, and graft-versus-host disease. We found that topical application of rhIL-2 can effectively relieve pain and improve the condition of oral mucosa for PV patients. Studies have shown that IL-2 selectively modulates CD4+ T cell subsets and increases the amounts and function of regulatory T cells. Moreover, IL-2 plays an important role in the proliferation of fibroblasts and wound healing. These evidences provide us the theoretical basis to explore the potential mechanism of rhIL-2 in treatment of mucosal damage of patients with PV.

Design of Study: This is a randomized, controlled, double-blind, multicenter clinical trial to assess the safety and short-term efficacy of rhIL-2 for oral erosion in patients with pemphigus.

Methods: rhIL-2 oral gargle combined with the standard dose of glucocorticoids (mucosal-dominant PV: prednisone 0.5 mg/kg/d, mucocutaneous PV: prednisone 1 mg/kg/d) will be applied to pemphigus patients meeting the inclusion criteria. The end points include clinical response and immunological changes, as well as safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 18 years and 70 years;
2. Patients definitely diagnosed with pemphigus vulgaris according to 'Diagnostic Criteria for Pemphigus Vulgaris (Autoimmune Disease Sub-Professional Committee of Dermatologist Branch of Chinese Medical Doctor Association)'; or pemphigus vulgaris has been diagnosed in the past.
3. Visible oral mucosa lesion due to pemphigus;
4. Mucosal-dominant PV or moderate mucocutaneous PV (PDAI score: 15-45);
5. Written informed consent was obtained, volunteer to participate in the project and complete as required.

Exclusion Criteria:

1. Patients with severe diseases of heart, brain, lungs, liver, kidney or blood system; patients experienced organ transplantation;
2. Patients with any acute severe infection such as pyemia and cellulitis, active tuberculosis, or an infection history of human immunodeficiency virus (HIV);
3. Patients with allergic skin diseases with obvious pruritus such as eczema or urticaria, blood routine examination show elevated eosinophils or have a clear history of allergy to rhIL-2;
4. Patients with persistent ventricular tachycardia, uncontrolled arrhythmias, chest pain with ECG changes, angina or myocardial infarction, cardiac tamponade;
5. Patients with nausea, vomiting, peptic ulcer or intestinal ischemia;
6. Patients with drug abuse, alcohol abuse, or mental disorders that are unable to cooperate or adhere to treatment;
7. Pregnant women, lactating women or women who are ready to conceive within 3 months;
8. Patients receiving treatment of immunosuppressants in the last 3 months;
9. Patients receiving continuous treatment of glucocorticoids with a dose of more than 0.75 mg/kg/d in the last 2 weeks;
10. Patients with oral fungal infection but don't receive antifungal therapy;
11. Participated in other clinical trials within 3 months before the screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The decline of the oral mucosa score of Pemphigus Disease Area Index (PDAI) after a 21-day treatment. | from baseline to 21 days treatment
  (PDAI score on Day 0 - PDAI score on Day 21)/PDAI score on Day 0 × 100%

SECONDARY OUTCOMES:
The decline of the oral mucosa score of Pemphigus Disease Area Index (PDAI) after a 7-, 14-, 28- and 42-day treatment, respectively. | from baseline to 7, 14, 28 and 42 days, respectively
  (PDAI score on Day 0 - PDAI score on Day N)/PDAI score on Day 0 × 100%
The decline of Oral Disease Severity Score (ODSS) after a 7-, 14-, 21-, 28- and 42-day treatment, respectively. | from baseline to 7, 14, 21, 28 and 42 days, respectively
  (ODSS on Day 0 - ODSS on Day N)/ODSS on Day 0 × 100%
The decline of oral mucosa Visual Analogue Scale(VAS) after a 7-, 14-, 21-, 28- and 42-day treatment, respectively. | from baseline to 7, 14, 21, 28 and 42 days, respectively
  (VAS on Day 0 - VAS on Day N)/VAS on Day 0 × 100%
The decline of Physician's Global Assessment (PGA) score for oral mucosa damage after a 7-, 14-, 21-, 28- and 42-day treatment, respectively. | from baseline to 7, 14, 21, 28 and 42 days, respectively
  (PGA score on Day 0 - PGA score on Day N)/PGA score on Day 0 × 100%
The decline of sera autoantibodies titer after a 21- and 42-day treatment, respectively. | from baseline to 21 and 42 days, respectively
  The autoantibodies including anti-Dsg3 and anti-Dsg1 antibodies titer are detected by ELISA
The dose of glucocorticoids on Day 28 and Day 42, respectively. | 28 and 42 days
  prednisone (mg/d)
The percentage of patients receiving incremental dose of glucocorticoids, steroid pulse therapy, or combined with immunosuppressants/intravenous immunoglobulin(IVIG)/biological agents on Day 28 and Day 42, respectively. | 28 and 42 days
The percentage of patients from whose oral mucosa the fungal infection can be detected on Day 21 and Day 42. | 21 and 42 days
The change of white blood cell (WBC) counts on Day 21 and Day 42. | 21 and 42 days
  The unit of WBC: 10^9/L
The change of serum potassium level on Day 21 and Day 42. | 21 and 42 days
  The unit of serum potassium level: mmol/L
The change of fasting blood-glucose (FBS) level on Day 21 and Day 42. | 21 and 42 days
  The unit of FBS level: mmol/L
The change of serum albumin level on Day 21 and Day 42. | 21 and 42 days
  The unit of serum albumin level: g/L
The safety evaluation about the drug adverse reactions throughout the entire study process. | through study completion, an average of 42 days
  the adverse reactions of rhIL-2 include fever, shiver, muscular soreness, nausea, emesis, rash, capillary leak syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No